CLINICAL TRIAL: NCT01785875
Title: A Multicenter Single-arm Extension Study to Describe the Long-term Efficacy and Safety of AMG 416 in the Treatment of Secondary Hyperparathyroidism in Subjects With Chronic Kidney Disease on Hemodialysis
Brief Title: Extension Study of Etelcalcetide in the Treatment of Secondary Hyperparathyroidism (SHPT) in Patients With Chronic Kidney Disease (CKD) on Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120231; KAI-4169-008 (Other: KAI Pharmaceuticals, Inc (wholly owned subsidiary of Amgen Inc.)); 2012-002808-41 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Hyperparathyroidism, Secondary
Keywords: Secondary Hyperparathyroidism (SHPT), chronic kidney disease (CKD), hemodialysis, parathyroid hormone (PTH), hypocalcemia, bone and mineral metabolism
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic; Hypocalcemia | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Etelcalcetide (Experimental): Participants received etelcalcetide at a starting dose of 5 mg three times a week (TIW) for up to 52 weeks. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered by bolus injection into the venous line of the dialysis circuit at the end of hemodialysis treatment, and prior to or during rinse-back with each hemodialysis session (ie, 3 times per week).
  Other Names: AMG 416

SUMMARY:
This study is designed to describe the long-term safety and efficacy of etelcalcetide (AMG 416) for the treatment of SHPT in adults with CKD on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.
* Subject must complete the treatment and follow-up period, or have been discontinued for rising intact parathyroid hormone (iPTH), from an AMG 416 phase 3 parent study prior to the start of dosing in this study: 20120229 (NCT01785849), 20120230 (NCT01788046), or 20120359 (NCT01932970).
* Subject agrees to not participate in another study of an investigational agent during the study.
* Other Inclusion Criteria may apply

Exclusion Criteria:

* Currently receiving treatment in another investigational device or drug study.
* Currently receiving other investigational procedures while participating in this study.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Subject has an unstable medical condition based on medical history, physical examination, and routine laboratory tests, or is otherwise unstable in the judgment of the Investigator.

Other Exclusion Criteria may apply

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 891 (Actual)
Dates: Start 2013-07-31 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (178):
- United States (89):
  - Research Site, Birmingham, Alabama
  - Research Site, Pine Bluff, Arkansas
  - Research Site, Azusa, California
  - Research Site, Bakersfield, California
  - Research Site, Chula Vista, California
  - Research Site, Cudahy, California
  - Research Site, Fairfield, California
  - Research Site, Glendale, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site, Northridge, California
  - Research Site, Norwalk, California
  - Research Site, Ontario, California
  - Research Site, Riverside, California
  - Research Site, San Gabriel, California
  - Research Site, Simi Valley, California
  - Research Site, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Stamford, Connecticut
  - Research Site, Coral Springs, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Ocala, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pinecrest, Florida
  - Research Site, Tampa, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Evanston, Illinois
  - Research Site, Gurnee, Illinois
  - Research Site, Merrillville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Wichita, Kansas
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Lafayette, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Brookhaven, Mississippi
  - Research Site, Columbus, Mississippi
  - Research Site, Gulfport, Mississippi
  - Research Site, Tupelo, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Eatontown, New Jersey
  - Research Site, Brooklyn, New York
  - Research Site, Great Neck, New York
  - Research Site, Orchard Park, New York
  - Research Site, Ridgewood, New York
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Yonkers, New York
  - Research Site, Carrboro, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Columbia, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Austin, Texas
  - Research Site, Edinburg, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Grand Prairie, Texas
  - Research Site, Houston, Texas
  - Research Site, Lubbock, Texas
  - Research Site, Mansfield, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Mechanicsville, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Bluefield, West Virginia
- Australia (7):
  - Research Site, Liverpool, New South Wales
  - Research Site, St Leonards, New South Wales
  - Research Site, Westmead, New South Wales
  - Research Site, Brisbane, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Clayton, Victoria
  - Research Site, Parkville, Victoria
- Austria (3):
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (8):
  - Research Site, Aalst
  - Research Site, Baudour
  - Research Site, Bonheiden
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
  - Research Site, Tournai
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Brampton, Ontario
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
- Czechia (7):
  - Research Site, Hradec Králové
  - Research Site, Nový Jičín
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Praha 4 - Nusle
  - Research Site, Slavkov u Brna
  - Research Site, Ústí nad Orlicí
- France (7):
  - Research Site, Bordeaux
  - Research Site, Caen
  - Research Site, La Tronche
  - Research Site, Marseille
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Saint-Ouen
- Germany (4):
  - Research Site, Berlin
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Villingen-Schwenningen
- Hungary (9):
  - Research Site, Baja
  - Research Site, Budapest
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Zalaegerszeg
- Israel (7):
  - Research Site, Ashkelon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
  - Research Site, Ẕerifin
- Italy (5):
  - Research Site, Ancona
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Pavia
  - Research Site, Verona
- Netherlands (4):
  - Research Site, Amsterdam
  - Research Site, Enschede
  - Research Site, Rotterdam
  - Research Site, Venlo
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Golub-Dobrzyń
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Rybnik
  - Research Site, Warsaw
  - Research Site, Zamość
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Spain (5):
  - Research Site, Córdoba, Andalusia
  - Research Site, Santander, Cantabria
  - Research Site, Barcelona, Catalonia
  - Research Site, Majadahonda, Madrid
  - Research Site, Madrid
- Sweden (3):
  - Research Site, Karlstad
  - Research Site, Stockholm
  - Research Site, Uppsala
- United Kingdom (5):
  - Research Site, Cambridge
  - Research Site, Coventry
  - Research Site, London
  - Research Site, Nottingham
  - Research Site, Sheffield

REFERENCES:
- [Background] Block GA, Chertow GM, Sullivan JT, Deng H, Mather O, Tomlin H, Serenko M. An integrated analysis of safety and tolerability of etelcalcetide in patients receiving hemodialysis with secondary hyperparathyroidism. PLoS One. 2019 Mar 15;14(3):e0213774. doi: 10.1371/journal.pone.0213774. eCollection 2019. PMID 30875390
- [Derived] Bushinsky DA, Chertow GM, Cheng S, Deng H, Kopyt N, Martin KJ, Rastogi A, Urena-Torres P, Vervloet M, Block GA. One-year safety and efficacy of intravenous etelcalcetide in patients on hemodialysis with secondary hyperparathyroidism. Nephrol Dial Transplant. 2020 Oct 1;35(10):1769-1778. doi: 10.1093/ndt/gfz039. PMID 30859218
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-arm study was conducted at 205 centers in the US, Canada, Europe, Israel, Russian Federation and Australia. Participants were enrolled from 31 July 2013 to 9 June 2014.
  Participants who rolled over into another single-arm extension study 20130213 (NCT02102204) are reported as discontinuing the study due to protocol specified criteria.
Pre-assignment Details: This extension study enrolled participants from 1 of 3 parent studies: 20120229 (NCT01785849), 20120230 (NCT01788046), or 20120359 (NCT01932970). In Studies 20120229 and 20120230, patients received either placebo or etelcalcetide 3 times a week (TIW) for up to 26 weeks; In Study 20120359, patients received 5 mg etelcalcetide TIW for 4 weeks.
Groups:
- 20120229 / 20120230 Placebo: Participants who received placebo in parent study 20120229 or 20120230 received etelcalcetide at a starting dose of 5 mg three times a week (TIW) for up to 52 weeks in the extension study. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
- 20120229 / 20120230 Etelcalcetide: Participants who received etelcalcetide in parent study 20120229 or 20120230 received etelcalcetide at a starting dose of 5 mg TIW for up to 52 weeks in the extension study. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
- 20120359 Etelcalcetide: Participants who received etelcalcetide in parent study 20120359 received etelcalcetide at a starting dose of 5 mg TIW for up to 52 weeks in the extension study. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
Period: Overall Study
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide
Started | 384 | 384 | 123
Received Etelcalcetide | 383 | 384 | 123
Completed | 90 (Completed etelcalcetide and the 30-day safety follow-up period) | 95 (Completed etelcalcetide and the 30-day safety follow-up period) | 16 (Completed etelcalcetide and the 30-day safety follow-up period)
Not Completed | 294 | 289 | 107
Not completed — Withdrawal by Subject | 41 | 34 | 36
Not completed — Lost to Follow-up | 19 | 22 | 6
Not completed — Death | 27 | 16 | 7
Not completed — Sponsor Decision | 0 | 2 | 0
Not completed — Protocol Specified Criteria | 207 | 214 | 55
Not completed — Missing | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Etelcalcetide: All participants received etelcalcetide at a starting dose of 5 mg TIW for up to 52 weeks during the extension study. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
Arm/Group | Etelcalcetide
Number analyzed (Participants) | 891
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (14.4)
Age, Customized [Number; unit: participants]
  < 65 years | 577
  ≥ 65 years | 314
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 341
  Male | 550
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 29
  Black (or African American) | 270
  Native Hawaiian or Other Pacific Islander | 12
  White | 567
  Other | 12
Ethnicity [Number; unit: participants]
  Hispanic/Latino | 122
  Not Hispanic/Latino | 769
Parathyroid Hormone (PTH) Level [Number; unit: participants]
  < 600 pg/mL | 405
  600 - ≤ 1000 pg/mL | 221
  > 1000 pg/mL | 228
  Missing | 37
PTH Concentration [Mean (Standard Deviation); unit: pg/mL] — Data available for 854 participants
  pg/mL | 769.5 (574.4)
Corrected Calcium [Mean (Standard Deviation); unit: mg/dL] — Data available for 889 participants
  mg/dL | 9.67 (0.68)
Phosphorus [Mean (Standard Deviation); unit: mg/dL] — Data available for 887 participants
  mg/dL | 5.63 (1.75)
Corrected Calcium Phosphorus Product (cCa x P) [Mean (Standard Deviation); unit: mg²/dL²] — Data available for 887 participants
  mg²/dL² | 54.36 (17.17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-related adverse events are those the investigator indicated as having a reasonable possibility of having been caused by etelcalcetide. A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria: • fatal • life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • congenital anomaly/birth defect • other medically important serious event.
Time Frame: From first dose until 30 days after last dose; the treatment period was 52 weeks.
Population: All participants who received at least 1 dose of etelcalcetide.
Measure: Number; unit: participants
Groups:
- Etelcalcetide Total: Participants received etelcalcetide at a starting dose of 5 mg three times a week (TIW) for up to 52 weeks. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 383 | 384 | 123 | 890
participants
  Any adverse event | 354 | 337 | 108 | 799
  Serious adverse events | 161 | 142 | 53 | 356
  Treatment-related adverse events | 215 | 141 | 36 | 392
  Treatment-related serious adverse events | 6 | 5 | 2 | 13
  AEs leading to discontinuation of etelcalcetide | 22 | 11 | 8 | 41
  Fatal adverse events | 27 | 16 | 8 | 51

2. Primary Outcome: Number of Participants With Shift in Laboratory Values From Baseline Grade 0 or 1 to Post-baseline Grade 3 or 4
Description: Laboratory toxicity grading was based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, where Grade 0 represents values in the normal range and grade 4 represents values with life-threatening consequences and urgent intervention indicated.
Time Frame: 52 weeks
Population: All participants who received at least 1 dose of etelcalcetide.
Measure: Number; unit: participants
Arm/Group | Etelcalcetide Total
Number analyzed (Participants) | 890
participants
  Alanine aminotransferase increase | 1
  Albumin decrease | 9
  Alkaline phosphatase increase | 2
  Aspartate aminotransferase increase | 3
  Bilirubin increase | 1
  Calcium (corrected) decrease | 51
  Calcium (corrected) increase | 8
  Phosphorus decrease | 77
  Potassium decrease | 9
  Potassium increase | 69
  Hemoglobin decrease | 4
  Hemoglobin increase | 1

3. Primary Outcome: Number of Participants Who Developed Anti-etelcalcetide Antibodies
Description: A validated dual flow-cell biosensor immunoassay was used to detect antibodies capable of binding etelcalcetide. The number of participants with a negative or no result at baseline and positive binding antibodies at any time post-baseline is reported.
Time Frame: Baseline, Week 12, Week 24, Week 36, Week 53, the 30-day follow-up visit
Population: Participants who received at least 1 dose of etelcalcetide and with a post-baseline antibody result.
Measure: Number; unit: participants
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 369 | 384 | 123 | 876
participants | 10 | 15 | 2 | 27

4. Secondary Outcome: Percentage of Participants With > 30% Reduction From Baseline in PTH During the Efficacy Assessment Phase
Description: The efficacy assessment phase (EAP) is defined as the last 6 weeks before ending treatment, which was only for participants who completed a minimum of 8 weeks of treatment with etelcalcetide. If multiple assessments were available during the EAP, values were averaged.
Time Frame: Baseline and the efficacy assessment phase, defined as the last 6 weeks prior to ending treatment for participants who completed a minimum of 8 weeks of treatment (weeks 46-52 for participants who completed 52 weeks of treatment)
Population: Participants with pre-dialysis PTH assessment at baseline and during the EAP who completed a minimum of 8 weeks of treatment with etelcalcetide.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 341 | 332 | 106 | 779
percentage of participants | 81.2 [76.7 to 85.2] | 54.5 [49.0 to 60.0] | 65.1 [55.2 to 74.1] | 67.7 [64.2 to 70.9]

5. Secondary Outcome: Percentage of Participants With > 30% Reduction From Baseline in PTH During the EAP12
Description: The efficacy assessment phase at 12 months (EAP12) was defined as the period from week 46 to 53 (inclusive). If multiple assessments were available during the EAP12, values were averaged.
Time Frame: Baseline and the efficacy assessment phase at month 12 (weeks 46-53)
Population: Participants with pre-dialysis PTH assessment at baseline and during EAP12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 302 | 300 | 74 | 676
percentage of participants | 82.5 [77.7 to 86.6] | 53.3 [47.5 to 59.1] | 63.5 [51.5 to 74.4] | 67.5 [63.8 to 71.0]

6. Secondary Outcome: Percentage of Participants With PTH ≤ 300 pg/mL During the EAP
Time Frame: Baseline and the efficacy assessment phase
Population: Participants with predialysis PTH assessment during the EAP who completed a minimum of 8 weeks of treatment with etelcalcetide
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 352 | 355 | 108 | 815
percentage of participants | 55.7 [50.3 to 60.9] | 59.7 [54.4 to 64.9] | 54.6 [44.8 to 64.2] | 57.3 [53.8 to 60.7]

7. Secondary Outcome: Percentage of Participants With PTH ≤ 300 pg/mL During the EAP12
Time Frame: Week 46 to 53
Population: Participants with predialysis PTH assessment during the EAP12
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 312 | 321 | 75 | 708
percentage of participants | 54.8 [49.1 to 60.4] | 61.1 [55.5 to 66.4] | 42.7 [31.3 to 54.6] | 56.4 [52.6 to 60.0]

8. Secondary Outcome: Percent Change From Baseline in Mean PTH During the EAP
Time Frame: Baseline and the efficacy assessment phase
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 341 | 332 | 106 | 779
percent change | -54.55 (2.12) | 3.92 (8.68) | -28.40 (6.96) | -26.07 (4.04)

9. Secondary Outcome: Percent Change From Baseline in Mean PTH During the EAP12
Time Frame: Baseline and the efficacy assessment phase at month 12 (weeks 46-53)
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 302 | 300 | 74 | 676
percent change | -55.41 (2.20) | 4.78 (9.62) | -27.05 (7.57) | -25.59 (4.59)

10. Secondary Outcome: Percent Change From Baseline in Mean Corrected Calcium During the EAP
Time Frame: Baseline and the efficacy assessment phase
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 352 | 352 | 103 | 807
percent change | -10.01 (0.52) | -6.74 (0.47) | -8.65 (1.04) | -8.41 (0.34)

11. Secondary Outcome: Percent Change From Baseline in Mean Corrected Calcium During the EAP12
Time Frame: Baseline and the efficacy assessment phase at month 12 (weeks 46-53)
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 310 | 319 | 75 | 704
percent change | -9.76 (0.52) | -6.43 (0.45) | -9.73 (1.14) | -8.25 (0.34)

12. Secondary Outcome: Percent Change From Baseline in Mean Corrected Calcium Phosphorus Product During the EAP
Time Frame: Baseline and the efficacy assessment phase
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 342 | 345 | 99 | 786
percent change | -15.26 (1.58) | -10.41 (1.61) | -6.58 (4.28) | -12.04 (1.13)

13. Secondary Outcome: Percent Change From Baseline in Mean Corrected Calcium Phosphorus Product During the EAP12
Time Frame: Baseline and the efficacy assessment phase at month 12 (weeks 46-53)
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 309 | 317 | 75 | 701
percent change | -15.30 (1.53) | -9.78 (1.62) | -7.29 (4.82) | -11.95 (1.13)

14. Secondary Outcome: Percent Change From Baseline in Mean Phosphorus During the EAP
Time Frame: Baseline and the efficacy assessment phase
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 343 | 348 | 105 | 796
percent change | -5.71 (1.71) | -3.50 (1.68) | 2.82 (4.56) | -3.62 (1.20)

15. Secondary Outcome: Percent Change From Baseline in Mean Phosphorus During the EAP12
Time Frame: Baseline and the efficacy assessment phase at month 12 (weeks 46-53)
Population: Participants with available data
Measure: Mean (Standard Error); unit: percent change
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 309 | 319 | 75 | 703
percent change | -5.87 (1.65) | -3.06 (1.73) | 3.53 (5.46) | -3.59 (1.22)

16. Primary Outcome: Change From Baseline in Blood Pressure
Description: Blood pressure (BP) values were taken post-hemodialysis assessments.
Time Frame: Baseline and Weeks 24 and 48
Population: Participants who received at least 1 dose of etelcalcetide and with available data at each time point (indicated by n)
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Etelcalcetide Total
Number analyzed (Participants) | 383 | 384 | 123 | 890
mmHg
  Systolic BP Week 24 (n = 329, 342, 104, 775) | 4.0 (1.5) | 4.5 (1.4) | -5.5 (2.8) | 2.9 (1.0)
  Systolic BP Week 48 (n = 305, 317, 74, 696) | 3.5 (1.6) | 6.5 (1.5) | -6.8 (3.0) | 3.8 (1.0)
  Diastolic BP Week 24 (n = 329, 343, 104, 776) | 2.2 (0.8) | 1.2 (0.9) | -5.1 (1.5) | 0.8 (0.6)
  Diastolic BP Week 48 (n = 305, 317, 74, 696) | 1.1 (0.9) | 0.8 (0.9) | -2.6 (1.7) | 0.6 (0.6)

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after last dose; the treatment period was 52 weeks.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Total: Participants received etelcalcetide at a starting dose of 5 mg three times a week (TIW) for up to 52 weeks. Etelcalcetide dose could be increased at weeks 5, 9, 17, 25, 33, 41, and 49 to a maximum dose of 15 mg to achieve predialysis serum parathyroid hormone levels ≤ 300 pg/mL.
Arm/Group | 20120229 / 20120230 Placebo | 20120229 / 20120230 Etelcalcetide | 20120359 Etelcalcetide | Total
Serious Adverse Events (participants affected / at risk) | 161/383 | 142/384 | 53/123 | 356/890
Other Adverse Events (participants affected / at risk) | 289/383 | 249/384 | 75/123 | 613/890
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20120229 / 20120230 Placebo (N=383) | 20120229 / 20120230 Etelcalcetide (N=384) | 20120359 Etelcalcetide (N=123) | Total (N=890)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 2 | 6
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 3 | 0 | 1 | 4
Acute myocardial infarction (Cardiac disorders) | 5 | 6 | 0 | 11
Angina pectoris (Cardiac disorders) | 2 | 3 | 2 | 7
Angina unstable (Cardiac disorders) | 1 | 1 | 0 | 2
Aortic valve disease (Cardiac disorders) | 1 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 9 | 4 | 0 | 13
Atrial flutter (Cardiac disorders) | 1 | 1 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 1 | 3
Bradycardia (Cardiac disorders) | 2 | 2 | 1 | 5
Cardiac arrest (Cardiac disorders) | 6 | 2 | 4 | 12
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 3 | 0 | 5
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 8 | 7 | 3 | 18
Cardiac valve disease (Cardiac disorders) | 1 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 3 | 0 | 4
Cardiogenic shock (Cardiac disorders) | 1 | 1 | 0 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 6 | 0 | 9
Coronary artery stenosis (Cardiac disorders) | 3 | 0 | 0 | 3
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 4 | 1 | 7
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus node dysfunction (Cardiac disorders) | 0 | 2 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 2 | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0 | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 2 | 2 | 6
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0 | 3
Goitre (Endocrine disorders) | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 1
Lens dislocation (Eye disorders) | 1 | 0 | 0 | 1
Optic neuropathy (Eye disorders) | 1 | 0 | 0 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 1 | 7
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Anorectal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 0 | 4
Diverticular perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 4 | 4 | 10
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastrointestinal vascular malformation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Megacolon (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatic duct obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1 | 4
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 5
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 1
Asthenia (General disorders) | 2 | 2 | 1 | 5
Chest pain (General disorders) | 3 | 7 | 1 | 11
Device occlusion (General disorders) | 1 | 0 | 0 | 1
Drug resistance (General disorders) | 1 | 0 | 0 | 1
Haemorrhagic cyst (General disorders) | 0 | 1 | 0 | 1
Hyperthermia (General disorders) | 1 | 0 | 0 | 1
Hyperthermia malignant (General disorders) | 0 | 0 | 1 | 1
Hypothermia (General disorders) | 1 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 1 | 0 | 1
Non-cardiac chest pain (General disorders) | 6 | 5 | 1 | 12
Pyrexia (General disorders) | 2 | 2 | 3 | 7
Sudden death (General disorders) | 1 | 1 | 1 | 3
Thrombosis in device (General disorders) | 1 | 0 | 2 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 3 | 0 | 5
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 0 | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 1
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Acinetobacter infection (Infections and infestations) | 0 | 1 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 1 | 1 | 2 | 4
Bacteraemia (Infections and infestations) | 2 | 2 | 0 | 4
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Bacterial tracheitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 | 2
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 8 | 4 | 1 | 13
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 1 | 2
Device related sepsis (Infections and infestations) | 1 | 1 | 1 | 3
Diabetic gangrene (Infections and infestations) | 0 | 1 | 1 | 2
Diverticulitis (Infections and infestations) | 1 | 1 | 0 | 2
Endocarditis (Infections and infestations) | 1 | 0 | 0 | 1
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 1
Gangrene (Infections and infestations) | 0 | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 6 | 0 | 0 | 6
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Genital abscess (Infections and infestations) | 1 | 0 | 0 | 1
Graft infection (Infections and infestations) | 0 | 0 | 1 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 2
Infected skin ulcer (Infections and infestations) | 3 | 1 | 0 | 4
Infectious mononucleosis (Infections and infestations) | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 3 | 1 | 2 | 6
Intervertebral discitis (Infections and infestations) | 2 | 0 | 0 | 2
Localised infection (Infections and infestations) | 0 | 1 | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 2
Osteomyelitis (Infections and infestations) | 4 | 3 | 1 | 8
Osteomyelitis acute (Infections and infestations) | 1 | 0 | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1 | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 7 | 5 | 3 | 15
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 1
Renal cyst infection (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 10 | 2 | 3 | 15
Septic shock (Infections and infestations) | 3 | 1 | 2 | 6
Shunt infection (Infections and infestations) | 0 | 1 | 0 | 1
Skin infection (Infections and infestations) | 1 | 1 | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 2 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 4
Urosepsis (Infections and infestations) | 1 | 2 | 0 | 3
Viral infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection (Infections and infestations) | 2 | 0 | 0 | 2
Wound sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 7 | 6 | 0 | 13
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 3 | 4 | 1 | 8
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 4 | 6 | 0 | 10
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Coronary bypass thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Dialysis related complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 3
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Peripheral arterial reocclusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Splenic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Stoma site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 4
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 4 | 2 | 2 | 8
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1
Anticoagulation drug level below therapeutic (Investigations) | 1 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 2
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1
Hepatitis C antibody positive (Investigations) | 1 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 2
Troponin increased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 3 | 8 | 4 | 15
Hyperkalaemia (Metabolism and nutrition disorders) | 14 | 10 | 5 | 29
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 4 | 1 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 2 | 0 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 3 | 1 | 4
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 2
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 2
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1
Meralgia paraesthetica (Nervous system disorders) | 0 | 0 | 1 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2 | 0 | 2
Seizure (Nervous system disorders) | 3 | 1 | 0 | 4
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 6 | 2 | 3 | 11
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 0 | 2
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 2 | 1 | 3
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 1 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 6 | 0 | 2 | 8
Azotaemia (Renal and urinary disorders) | 2 | 2 | 0 | 4
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 2
Nephrosclerosis (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal cyst haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Pelvic haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 5
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 5
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 5 | 0 | 6
Vasculitic rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Arteriovenous graft (Surgical and medical procedures) | 0 | 1 | 0 | 1
Therapy cessation (Surgical and medical procedures) | 0 | 0 | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 2
Dry gangrene (Vascular disorders) | 1 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0 | 0 | 1
Haematoma (Vascular disorders) | 2 | 0 | 0 | 2
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 5 | 4 | 1 | 10
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1 | 2
Hypertensive emergency (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 5 | 4 | 2 | 11
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 1
Malignant hypertension (Vascular disorders) | 0 | 2 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 1 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1 | 1 | 4
Peripheral vascular disorder (Vascular disorders) | 2 | 4 | 0 | 6
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0 | 1
Steal syndrome (Vascular disorders) | 1 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20120229 / 20120230 Placebo (N=383) | 20120229 / 20120230 Etelcalcetide (N=384) | 20120359 Etelcalcetide (N=123) | Total (N=890)
Abdominal pain (Gastrointestinal disorders) | 22 | 12 | 3 | 37
Diarrhoea (Gastrointestinal disorders) | 41 | 46 | 8 | 95
Nausea (Gastrointestinal disorders) | 43 | 27 | 13 | 83
Vomiting (Gastrointestinal disorders) | 40 | 37 | 11 | 88
Bronchitis (Infections and infestations) | 20 | 6 | 2 | 28
Nasopharyngitis (Infections and infestations) | 19 | 21 | 3 | 43
Upper respiratory tract infection (Infections and infestations) | 20 | 14 | 20 | 54
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 22 | 27 | 8 | 57
Fall (Injury, poisoning and procedural complications) | 22 | 14 | 6 | 42
Procedural hypotension (Injury, poisoning and procedural complications) | 17 | 8 | 8 | 33
Blood calcium decreased (Investigations) | 226 | 129 | 30 | 385
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 18 | 10 | 47
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 20 | 4 | 50
Muscle spasms (Musculoskeletal and connective tissue disorders) | 36 | 33 | 10 | 79
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 23 | 6 | 45
Headache (Nervous system disorders) | 25 | 25 | 2 | 52
Anxiety (Psychiatric disorders) | 8 | 10 | 7 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 20 | 13 | 54
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 17 | 5 | 46
Hypertension (Vascular disorders) | 30 | 18 | 10 | 58
Hypotension (Vascular disorders) | 36 | 25 | 5 | 66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.